CLINICAL TRIAL: NCT00868335
Title: Cervical Spine; Movement Before and After Anterior Cervical Discectomy, With or Without an Activ-C Cervical Disc Prosthesis.
Brief Title: Cervical Spine; Movement Before and After Anterior Cervical Discectomy, With or Without a Cervical Disc Prosthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: B. Braun/Aesculap Spine (Unknown)
Responsible Party: Principal Investigator, Toon Boselie, MD, Maastricht University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CWK-Tracking01
Record Dates: First submitted 2009-03-23; First posted 2009-03-24 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Diskectomy; Intervertebral Disk Displacement
Keywords: Cervical degenerative disc disease; Anterior cervical discectomy; Cervical disc prosthesis; Activ-C; Mobility; Movement
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Anterior cervical discectomy, no disc prosthesis
  Interventions: Procedure: Anterior cervical discectomy
- 2 (Experimental): Anterior cervical discectomy, with disc prosthesis
  Interventions: Device: Activ C disc prosthesis; Procedure: Anterior cervical discectomy

INTERVENTIONS:
Device: Activ C disc prosthesis — cervical disc prosthesis
  Other Names: Activ C cervical disc prosthesis, B.Braun/Aesculap Spine
  Arms: 2
Procedure: Anterior cervical discectomy — Removal of protruding cervical disc through an anterior approach

SUMMARY:
The purpose of this study is to find out if use of a cervical disc prosthesis in the treatment of a cervical disc herniation preserves or restores normal mobility and movement in the cervical spine.

DETAILED DESCRIPTION:
Intractable nerve pain to the arm caused by a cervical disc herniation is typically treated by removal of the protruding disc through an operation. Fusion of the discs follows in about 70% of cases.

Adjacent disc disease (ADD), symptomatic degenerative changes in the levels adjacent to the operated level is regarded as a late complication. Fusion at the operated level is thought to contribute to this process due to compensative increased mobility and stress on the adjacent segments.

Keeping the operated segment mobile through the use of a cervical disc prosthesis possibly prevents ADD.

We hypothesize that use of a cervical disc prosthesis preserves or restores normal mobility to the cervical spine. To test this hypothesis subjects are randomised in a group receiving a standard anterior cervical discectomy, and a group receiving a standard discectomy with placement of a cervical disc prosthesis. Digital X-ray cinematographic videos are made of a flexion/extension movement. The videos will be analyzed manually and through a newly designed automated program, to check for mobility and order of movement.

ELIGIBILITY:
Inclusion Criteria:

* indication for anterior cervical discectomy
* monoradicular syndrome caused by compression at C5-6 or C6-7
* monosegmental disease on MRI
* able to actively perform flexion/extension movement
* segmental mobility on the afflicted level >2 degrees of rotation
* informed consent

Exclusion Criteria:

* previous operative interventions on the cervical spine
* multiple segments afflicted
* positive L'Hermittes sing
* Active infection
* Immature bone
* Tumorous processes in the cervical region
* Previous radiation therapy in the cervical region
* Pregnancy
* Cervical myelopathy
* not able to speak Dutch

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2007-12; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Order of movement | baseline, 3 months, 12 months
Segmental mobility | Baseline, 3 months, 12 months

SECONDARY OUTCOMES:
Treatment of symptoms (pain, neurological assessment) | Baseline, 3 months, 12 months
Influence on subjects functioning (social, work) | Baseline, 3 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: H van Santbrink, MD, PhD, Principal Investigator — Department of Neurosurgery, Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Boselie TF, van Mameren H, de Bie RA, van Santbrink H. Cervical spine kinematics after anterior cervical discectomy with or without implantation of a mobile cervical disc prosthesis; an RCT. BMC Musculoskelet Disord. 2015 Feb 21;16:34. doi: 10.1186/s12891-015-0479-4. PMID 25887569